CLINICAL TRIAL: NCT03665259
Title: Effects of Preoxygenation With Lower Inspiratory Oxygen Fraction During Induction of Anesthesia
Brief Title: Lower Inspiratory Oxygen Fraction for Preoxygenation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Significantly increased incidence of primary endpoint in the FiO2 60% group
Sponsor: E-DA Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EMRP15107N
Record Dates: First submitted 2018-09-02; First posted 2018-09-11 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2018-09

CONDITIONS: Intraoperative Complications; Respiratory Complication; Oxygen Toxicity; Oxygen Deficiency; Anesthesia
Keywords: Oxygen; Perioperative medicine; General anesthesia; Preoxygenation
MeSH Terms: conditions — Intraoperative Complications; Hypoxia

STUDY DESIGN:
Intervention Model Description: Group 1: pre-oxygenation with 100% oxygen during induction of anesthesia Group 2: pre-oxygenation with 60% oxygen during induction of anesthesia
Who Masked: Participant, Outcomes Assessor
Masking Description: The anesthetist who in-charge of the induction of anesthesia is aware of the treatment oxygen concentration.
  The patient is unaware of oxygen concentration during the induction of anesthesia.
  The outcomes assessors is unaware of the concentration of oxygen treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pure oxygen group (Active Comparator): The patients receive 100% oxygen therapy during the induction phase of induction
  Interventions: Procedure: Pure oxygen group
- Lower oxygen group (Experimental): The patients received 60% oxygen therapy during the induction phase of induction
  Interventions: Procedure: Lower oxygen group

INTERVENTIONS:
Procedure: Pure oxygen group — pre-oxygenation with 100% oxygen during induction of anesthesia
  Arms: Pure oxygen group
Procedure: Lower oxygen group — Pre-oxygenation with 60% oxygen during induction of anesthesia
  Arms: Lower oxygen group

SUMMARY:
During the induction period of general anesthesia, surgical patients are inevitably experienced a short period of apnea for endotracheal intubation or other airway manipulation. In order to minimize the risks of hypoxemia during the establishment of artificial airway, pure oxygen (FiO2=100%) is commonly applied to the patients throughout the preoxygenation and induction period. However, high concentration of oxygen therapy has been shown to result in hyperoxemia and substantial oxygen exposure during perioperative period or critical care. There is currently no clinical evidence indicating that preoxygenation with a lower oxygen partial pressure (such as FiO2=60%) during the induction of anesthesia increases the incidence of hypoxemia or other complications. The findings of this proposed clinical study may provide fundamental evidence for the use of different oxygen concentrations in clinical anesthesia during the induction period, and determine the effects of inspired oxygen concentrations on the general postoperative outcomes during general anesthesia.

DETAILED DESCRIPTION:
The administration of 100% oxygen for 3-5 minutes may replace the nitrogen content in the lung cavity (de-nitrogenation) with higher alveolar concentrations of oxygen (greater then 95%). Elevation of oxygen reserve in the lung and oxygen partial pressure in the blood circulation may thus delay the development of hypoxemia (oxygen desaturation; defined as the tissue oxygen saturation below 90%) up to 10 minutes after apnea.

On the other hand, there is currently no clinical evidence indicating that preoxygenation with lower oxygen partial pressures (i.e. FiO2= 50-60%) during the induction of anesthesia increases the incidence of hypoxemia or other complications. Most recently, two elegant large-scale clinical trials reported that the supplement of oxygen to patients with acute myocardial infarction or acute ischemic stroke did not provide any clinically beneficial effects in the prognosis of diseases. The results of these two important trials did not support the routine supplement of oxygen in these acute diseases. In addition, high concentrations of oxygen therapy are potentially deleterious, as oxygen toxicity may result in direct tracheobronchial and alveolar damage, absorption atelectasis (lung tissue collapse) and central nervous system toxicity. In cellular levels, hyperoxia increases the production of reactive oxygen species, such as the superoxide anion, the hydroxyl radical, and hydrogen peroxide, which in turn may cause cellular apoptosis and inflammatory response. Therefore, oxygen therapy in clinical settings has been recognized as a two-edged sword and excessive oxygen supplement should be guided closely for its potential toxicity.

Currently, there is no clinical evidence that supports the routine administration of 100% oxygen prior to intubation is essential or beneficial. In the contrary, it also remains undetermined if lower fractions of inspiratory oxygen during the induction period of anesthesia may attenuate lung injury or other cellular damage derived from the oxygen toxicity. Therefore, the findings of this proposed clinical study may provide fundamental evidence for the use of different oxygen concentrations in clinical anesthesia during the induction period, and determine the effects of inspiratory oxygen concentrations on the general postoperative outcomes after general anesthesia.

This is a randomized, open-label, observer-blind and non-inferiority clinical trial.

The research model of study is two-group parallel interventional study. The control group is preoxygenation with 100% oxygen during the induction phase of anesthesia; the experimental group is preoxygenation with 60% oxygen during the induction phase of anesthesia. The anesthetists in-charge are not blinded to the concentrations of oxygen use during induction of anesthesia, but the persons who collected study data will be unaware of the treatment. Block randomization will be generated using a generator software and the assignment of treatment will be sealed in the envelops.

This study anticipates in enrolling 1500 participants.

ELIGIBILITY:
Inclusion Criteria:

1. A patient who is scheduled for an elective surgery and required for general anesthesia with endotracheal intubation.
2. Age of the patient is between 20 and 65 years old.
3. Patient's American Society of Anesthesiologists (ASA) Physical Status is I- III.

Exclusion Criteria:

Patients who:

1. Have difficult airway for ventilation or intubation.
2. Have severe lung disease (including any acute respiratory infection).
3. Had past history of coronary artery disease or myocardial infarction.
4. Have severe heart failure (NYHA Fc ≥III).
5. Have liver cirrhosis (Child-Pugh's score ≥B).
6. Have acute or chronic kidney disease (Creatinine ≥2 mg/dl).
7. Have severe anemia (hemoglobin ≤8 mg /dl).
8. Have a body mass index (BMI) ≥35.
9. Are currently pregnant.
10. Have inadequate fasting time, intestinal obstruction or severe gastroesophageal reflux.
11. Scheduled for an emergency surgery, cardiac surgery, craniotomy, or pulmonary surgery.
12. Have mental incapacitant, confusion, dementia, mental retardation, or are unable to complete the consent independently.
13. Refuse to participate in this study.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Incidence of hypoxemia | Within 30 minutes after induction of anesthesia
  The definition of hypoxemia is the measurement of peripheral oxygen saturation (sPO2) lower than < 92%. Induction phase of anesthesia is defined as the time frame from preoxygenation before intravenous administration of anesthetics to successful establishment of an endotracheal tube.

SECONDARY OUTCOMES:
Development of acute respiratory distress syndrome (ARDS) | Within 7 days after surgery
  ARDS is defined as any calculated PaO2/FiO2 less than 300mmHg with radiographic evidence of bilateral lung infiltration in the absence of left heart failure
Development of atelectasis | Within 7 days after surgery
  Atelectasis is defined as partial or complete collapse of lung lobe(s) on chest radiography
Development of pneumonia | Within 7 days after surgery
  Pneumonia is defined as acute infection of lung parenchyma
Development of surgical site infection (SSI) | Within 7 days after surgery
  SSI is defined as infection arising from surgical incision
Development of severe postoperative pain | Within 7 days after surgery
  Severe postoperative pain is defined as visual analogue scale (VAS) >4 despite of administration of analgesics. VAS is defined as a straight line with the endpoints representing the extreme limits of pain; "no pain at all= 0" and "pain as bad as it could be= 10"
Length of hospital stay (LOS) | Within 7 days after surgery
  LOS is defined as day(s) of hospitalization after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Chen-Fuh Lam, MD, PhD, Principal Investigator — E-DA Hospital
Locations (1):
- E-Da Hospital, Yanchao, Kaohsiung, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-11-20): https://cdn.clinicaltrials.gov/large-docs/59/NCT03665259/Prot_SAP_000.pdf
  • Informed Consent Form (2018-11-01): https://cdn.clinicaltrials.gov/large-docs/59/NCT03665259/ICF_001.pdf